CLINICAL TRIAL: NCT01620671
Title: The Feasibility of Fast-track Surgery for Perforated Peptic Ulcers. A Prospective Randomized Clinical Trial
Brief Title: Fast-track Surgery for Perforated Peptic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Gonenc, M.D., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTS-240310
Record Dates: First submitted 2012-06-11; First posted 2012-06-15 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Peptic Ulcer Perforation
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional surgery (Active Comparator): The patients who will have a conventional surgical treatment will be included.
  Interventions: Procedure: Surgical repair of perforated peptic ulcer
- Fast-track surgery (Active Comparator): The patients who will have fast-track surgery will be included.
  Interventions: Procedure: Surgical repair of perforated peptic ulcer

INTERVENTIONS:
Procedure: Surgical repair of perforated peptic ulcer — Perforated peptic ulcer located in the stomach and the duodenum will be repaired by either primary repair or omentoplasty.
  Arms: Conventional surgery
Procedure: Surgical repair of perforated peptic ulcer — Perforated peptic ulcer located in the stomach and the duodenum will be repaired by either primary repair or omentoplasty.
  Arms: Fast-track surgery

SUMMARY:
The concept of "enhanced recovery after surgery" has become increasingly popular in elective abdominal surgeries. Yet, the role of this concept has not been described in emergency procedures. Therefore, this study aimed to investigate the feasibility of fast-track surgery in patients with perforated peptic ulcer.

DETAILED DESCRIPTION:
The study is designed as a randomized, controlled clinical study. The patients with a preoperative diagnosis of perforated peptic ulcer will be recruited for the study. Among those, the patients with a definitive diagnosis of perforated peptic ulcer confirmed by surgical exploration will be included.

The patients will be randomized according to their protocol number given automatically by the registration system of the hospital during admission. The patients who have an odd protocol number will have conventional surgical protocol, and those who have an even protocol number will have fast-track surgery protocol.

The conventional surgical protocol for perforated peptic ulcers is composed of regular general anesthesia, postoperative pain control by intravenous analgesics, removal of nasogastric tube by the end of 48th postoperative hour, initiation of oral intake after clinical signs of active bowel movement is observed. Fast-track surgery protocol, however, is composed of general anesthesia with short-acting agents and the use of regional anesthesia if possible, removal of nasogastric tube during recovery from anesthesia, aggressive pain control, initiation of oral intake by the end of 48th postoperative hour.

All of the patients will be scheduled for control gastroscopy in the end of six weeks after surgery.

Primary end-point is the morbidity and mortality rate. Secondary end-points are length of hospital stay, readmission rate, endoscopic findings in control gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Perforated peptic ulcer located in the stomach or the duodenum

Exclusion Criteria:

* The patients who refuse to join the study or to sign the informed consent form
* The patients who are unable to understand and sign the informed consent form
* Age younger than 18
* The patients with a possibility of having trouble in communicating with or reaching the investigators during the first 6 weeks after surgery
* The patients who are considered as ASA class 4
* Shock on admission
* The patients who have serious negative factors for wound healing such as steroid usage, autoimmune diseases
* Pregnant
* Previous upper abdominal surgery
* The patients who are found to have a pathology other than perforated peptic ulcer during surgical exploration
* The patients who are found to have malignant ulcer during surgery or in postoperative period
* Concomitant bleeding peptic ulcers
* Peptic ulcer perforations with a diameter greater than 5 mm, which are not suitable for simple repair techniques
* Multiple perforated peptic ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The morbidity and mortality rate | First 6 weeks after surgery

SECONDARY OUTCOMES:
Length of hospital stay | An expected average of 5 days
  The participants will be followed for the duration of hospital stay.
Readmission rate | The period within the first 6 weeks after surgery
Endoscopic findings in control gastroscopy | At the end of 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Murat Gonenc, M.D., Principal Investigator — Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)